CLINICAL TRIAL: NCT03065907
Title: Timing of Low Vision Rehabilitation in Anti-VEGF Therapy: a Randomized, Controlled Trial
Brief Title: Timing of Low Vision Rehabilitation in Anti- Vascular Endothelial Growth Factor (VEGF) Therapy
Acronym: TRAVIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00141001
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Low Vision; Neovascular Age-related Macular Degeneration
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vision Rehabilitation Group 1 (Active Comparator): Vision rehabilitation assessment will be scheduled within 1 months of randomization; interventions will be scheduled and vision rehabilitation appointments will be scheduled accordingly.
  Interventions: Other: Vision rehabilitation
- Vision Rehabilitation Group 2 (Active Comparator): Vision rehabilitation assessment will be scheduled within 7 months of randomization; interventions will be scheduled and vision rehabilitation appointments will be scheduled accordingly.
  Interventions: Other: Vision rehabilitation

INTERVENTIONS:
Other: Vision rehabilitation — A service menu containing the minimum vision rehabilitation visits will be provided and assessed according to the participant's vision needs. Minimum vision rehabilitation visits include refraction, best-corrected visual acuity assessment, near vision, contrast sensitivity, central visual field test, education and consultation; rehabilitation visit will then be individualized.

SUMMARY:
The purpose of this research is to collect preliminary data in preparation for conducting a randomized clinical trial to determine the relative effectiveness of vision rehabilitation in improving overall visual ability (primary aim) and reducing depression (secondary aim) in patients receiving anti-VEGF therapy for neovascular age-related macular degeneration integrated over time.

DETAILED DESCRIPTION:
This is a pilot study to understand the feasibility of conducting a randomized, controlled trial regarding the timing for vision rehabilitation in patients receiving anti-VEGF therapy for neovascular age-related macular degeneration. Prior to initiating the clinical trial, the investigators must be assured that patients with loss in visual ability are willing to be randomized and amenable to deferring vision rehabilitation intervention. Although it is typical for patients receiving usual care to present for vision rehabilitation services years after the onset of anti-VEGF therapy, this manifestation may result from patients being unaware of the existence of vision rehabilitation services to enhance function and reduce depression. As part of the study recruitment, patients will be informed about vision rehabilitation care and, if suffering with difficulty performing everyday activities, they may be unwilling to defer vision rehabilitation. Additionally, the study design may not be feasible to answer the aim should patients in the delayed intervention arms suffer progressive loss in visual ability and seek vision rehabilitation services, resulting in a high drop-out rate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years old
* Primary diagnosis of neovascular age-related macular degeneration in the index eye or in both eyes if habitual visual acuity (HVA) is equivalent in both eyes
* HVA < 20/25 to ≥ 20/500 in the index eye
* Confirmed active anti-VEGF injections (a minimum of 2 injections in the past 3 months, a total of 8 injections maximum) in the index eye
* Full confrontational visual fields in the index eye
* Acknowledgement of having difficulty in visual ability function
* Visual ability estimates as measured by ≥ 2 goals identified on the Activity Inventory as important and with at least slight difficulty
* Telephone interview for cognitive status raw score is > 29
* Ability to return to clinic to participate in rehabilitation
* No prior experience with vision rehabilitation service

Exclusion Criteria:

* Other progressive ocular conditions likely to compromise VA during the study period or upcoming eye surgeries
* Anti-VEGF injections in the index eye 8 months prior to enrollment
* Unable to give written consent to the study
* Impaired hearing or cognitive ability that precludes telephone interviews
* Insufficient spoken English or reading ability to complete interviews and understand study materials

  * The index eye is defined as the eye with better HVA, or the eye with more anti-VEGF injections if both eyes are with the equivalent HVA

Ages: 50 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Consent rate | 2 months
  Consent rate of the approached participants

SECONDARY OUTCOMES:
Retention rate | 18 months
  Retention rate of the enrolled participants
Breaking of randomization in group 2 | 18 months
  Rate of participants crossing over to group 1 from group 2

CONTACTS AND LOCATIONS:
Overall Officials: Judith Goldstein, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States